CLINICAL TRIAL: NCT02064868
Title: A Multicenter, Prospective, Randomized, Open-label Study to Assess the Effect of Serelaxin Versus Standard of Care in Acute Heart Failure (AHF) Patients
Brief Title: Effect of Serelaxin Versus Standard of Care in Acute Heart Failure (AHF) Patients
Acronym: RELAX-AHF-EU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated based on results from pivotal adult AHF study CRLX030A2301
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRLX030A3301; 2013-002513-35 (EudraCT Number)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Acute Heart Failure (AHF)
Keywords: AHF,; RLX030,; SOC,; WHF,; RELAX-AHF-EU; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — serelaxin protein, human; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Serelaxin + Standard of Care (Experimental): Serelaxin (30 µg/kg/day) as continuous 48 hour intravenous infusion plus standard of care.
  Interventions: Drug: Serelaxin; Drug: Standard of Care
- Standard of Care (SOC) (Other): All patients were required to receive standard of care background heart failure (HF) management during the study, according to local guidelines/international standards. This treatment can include but is not limited to intravenous and/or oral diuretics, angiotensin-converting enzyme (ACE) inhibitors/angiotensin receptor antagonists, beta blockers and aldosterone receptor antagonists, etc.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Serelaxin — 30 µg/kg/day IV infusion
  Other Names: RLX030
  Arms: Serelaxin + Standard of Care
Drug: Standard of Care — This treatment can include but is not limited to intravenous and/or oral diuretics, angiotensin-converting enzyme (ACE) inhibitors/angiotensin receptor antagonists, beta blockers and aldosterone receptor antagonists, etc.

SUMMARY:
This was a multinational, multicenter, randomized, open-label study to confirm and expand the efficacy, safety and tolerability evidence of 48 hours intravenous infusion of serelaxin (30 micrograms/kg/day) when added to Standard of Care (SoC) in patients admitted to hospital for Acute Heart Failure (AHF).

DETAILED DESCRIPTION:
This study was aimed at generating clinical evidence, especially on the short term period (in-hospital and at 30 days) to complement existing and future serelaxin data sets in Acute Heart Failure (AHF).

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure ≥ 125 mmHg
* Admitted for Acute Heart Failure (AHF)
* Received intravenous furosemide (or equivalent) at any time between presentation and the start of screening
* eGFR on admission: ≥ 25 and ≤75 mL/min/1.73 m^2

Exclusion Criteria:

* Dyspnea (non-cardiac causes)
* T > 38.5°C
* Clinical evidence of acute coronary syndrome currently or within 30 days prior to enrollment.
* Significant left ventricular outflow obstruction, uncorrected, such as obstructive hypertrophic cardiomyopathy or severe aortic stenosis (i.e., aortic valve area <1.0 cm^2 or mean gradient >50 mmHg on prior or current echocardiogram), severe aortic regurgitation and severe mitral stenosis.
* AHF due to significant arrhythmias
* Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (does not include restrictive mitral filling patterns seen on Doppler echocardiographic assessments of diastolic function).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2666 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2017-03-26 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (313):
- Austria (6):
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Sankt Pölten
  - Novartis Investigative Site, Vienna
- Belgium (13):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Lodelinsart
  - Novartis Investigative Site, Mol
  - Novartis Investigative Site, Mons
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Ronse
  - Novartis Investigative Site, Turnhout
- Bulgaria (6):
  - Novartis Investigative Site, Gabrovo
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sliven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Veliko Tarnovo
- Croatia (2):
  - Novartis Investigative Site, Varaždin, HRV
  - Novartis Investigative Site, Zagreb
- Czechia (11):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Decin II, Czech Republic
  - Novartis Investigative Site, Karvina-Raj, Czech Republic
  - Novartis Investigative Site, Kroměříž, Czech Republic
  - Novartis Investigative Site, Mělník, Czech Republic
  - Novartis Investigative Site, Písek, Czech Republic
  - Novartis Investigative Site, Svitavy, Czech Republic
  - Novartis Investigative Site, Tábor, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Turku, Finland
- France (40):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Nancy, Cedex
  - Novartis Investigative Site, Abbeville
  - Novartis Investigative Site, Agen
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Belfort
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Chalon-sur-Saône
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Châteauroux
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Dunkirk
  - Novartis Investigative Site, La Seyne-sur-Mer
  - Novartis Investigative Site, Le Coudray
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lens
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lorient
  - Novartis Investigative Site, Metz
  - Novartis Investigative Site, Montauban
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Mulhouse
  - Novartis Investigative Site, Niort
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Orléans
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pau
  - Novartis Investigative Site, Périgueux
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Brieuc
  - Novartis Investigative Site, Saint-Michel-sur-Orge
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Troyes
  - Novartis Investigative Site, Vienne
- Germany (76):
  - Novartis Investigative Site, Flensburg, Schleswig-Holstein
  - Novartis Investigative Site, Arnstadt
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Baden-Baden
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bernburg
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Buchholz in der Nordheide
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dorsten
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düssledorf
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Eschwege
  - Novartis Investigative Site, Esslingen am Neckar
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Friesoythe
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Gotha
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Gütersloh
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heidenheim
  - Novartis Investigative Site, Hennigsdorf
  - Novartis Investigative Site, Herford
  - Novartis Investigative Site, Hoyerswerda
  - Novartis Investigative Site, Kaufbeuren
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Koeln-Nippes
  - Novartis Investigative Site, Langen
  - Novartis Investigative Site, Lemgo
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Marl
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neumünster
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Neustadt A.d. Aisch
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ribnitz-Damgarten
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rotenburg (Wümme)
  - Novartis Investigative Site, Schönebeck
  - Novartis Investigative Site, Schwabach
  - Novartis Investigative Site, Schwalmstadt
  - Novartis Investigative Site, Singen
  - Novartis Investigative Site, Soest
  - Novartis Investigative Site, Sonneberg
  - Novartis Investigative Site, Speyer
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stadtlohn
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Suhl
  - Novartis Investigative Site, Torgau
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Vechta
  - Novartis Investigative Site, Wesel
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Worms
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Wurzen
  - Novartis Investigative Site, Würzburg
- Greece (4):
  - Novartis Investigative Site, Alexandroupoli, Evros
  - Novartis Investigative Site, Voula, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Volos
- Hungary (10):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Kalocsa
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szolnok
- Novartis Investigative Site, Reykjavik, Iceland
- Italy (30):
  - Novartis Investigative Site, San Benedetto del Tronto, AP
  - Novartis Investigative Site, Arezzo, AR
  - Novartis Investigative Site, Acquaviva delle Fonti, BA
  - Novartis Investigative Site, Altamura, BA
  - Novartis Investigative Site, Cassano delle Murge, BA
  - Novartis Investigative Site, Treviglio, BG
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Lodi, LO
  - Novartis Investigative Site, Latina, LT
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Cernusco sul Naviglio, MI
  - Novartis Investigative Site, Legnano, MI
  - Novartis Investigative Site, Matera, Mount
  - Novartis Investigative Site, Piacenza, PC
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Scandiano, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Syracuse, SR
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Busto Arsizio, VA
  - Novartis Investigative Site, Chioggia, VE
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Vibo Valentia, VV
  - Novartis Investigative Site, Pozzuoli
- Novartis Investigative Site, Daugavpils, Latvia
- Lithuania (4):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Vilnius
- Poland (13):
  - Novartis Investigative Site, Krakow, POL
  - Novartis Investigative Site, Biłgoraj
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Grodzisk Mazowiecki
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lubin
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Oświęcim
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Tarnobrzeg
  - Novartis Investigative Site, Tarnów
  - Novartis Investigative Site, Wałbrzych
- Portugal (7):
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Barreiro
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Setúbal
  - Novartis Investigative Site, Vila Franca de Xira
- Romania (6):
  - Novartis Investigative Site, Bucharest, District 4
  - Novartis Investigative Site, Bucharest, Jud Cluj
  - Novartis Investigative Site, Craiova, Jud. Iasi
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Sibiu
  - Novartis Investigative Site, Târgovişte
- Russia (21):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Chita
  - Novartis Investigative Site, Gatchina
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Vladivostok
  - Novartis Investigative Site, Volgograd
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Zelenograd, Moscow Region
- Serbia (4):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Kamenica
  - Novartis Investigative Site, Niš
  - Novartis Investigative Site, Niška Banja
- Slovakia (6):
  - Novartis Investigative Site, Dunajská Streda, Slovak Republic
  - Novartis Investigative Site, Skalica, Slovak Republic
  - Novartis Investigative Site, Zvolen, Slovak Republic
  - Novartis Investigative Site, Brezno
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Trenčín
- Slovenia (4):
  - Novartis Investigative Site, Celje
  - Novartis Investigative Site, Jesenice
  - Novartis Investigative Site, Ljubljana
  - Novartis Investigative Site, Murska Sobota
- Spain (31):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Galdakano, Basque Country
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Soria, Castille and León
  - Novartis Investigative Site, Toledo, Castille-La Mancha
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, Cartagena, Murcia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Manises, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, León
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Murcia
  - Novartis Investigative Site, Zaragoza
- Switzerland (4):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Liestal
  - Novartis Investigative Site, Lugano
- United Kingdom (10):
  - Novartis Investigative Site, Durham, County Durham
  - Novartis Investigative Site, Dorchester, Dorset
  - Novartis Investigative Site, Peterborough, GBR
  - Novartis Investigative Site, Gateshead, Tyne and Wear
  - Novartis Investigative Site, Barnet
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Dundee
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Swindon

REFERENCES:
- [Derived] Grand J, Miger K, Sajadieh A, Kober L, Torp-Pedersen C, Ertl G, Lopez-Sendon J, Pietro Maggioni A, Teerlink JR, Sato N, Gimpelewicz C, Metra M, Holbro T, Nielsen OW. Blood Pressure Drops During Hospitalization for Acute Heart Failure Treated With Serelaxin: A Patient-Level Analysis of 4 Randomized Controlled Trials. Circ Heart Fail. 2022 Apr;15(4):e009199. doi: 10.1161/CIRCHEARTFAILURE.121.009199. Epub 2022 Feb 21. PMID 35184572
- [Derived] Grand J, Miger K, Sajadieh A, Kober L, Torp-Pedersen C, Ertl G, Lopez-Sendon J, Pietro Maggioni A, Teerlink JR, Sato N, Gimpelewicz C, Metra M, Holbro T, Nielsen OW. Systolic Blood Pressure and Outcome in Patients Admitted With Acute Heart Failure: An Analysis of Individual Patient Data From 4 Randomized Clinical Trials. J Am Heart Assoc. 2021 Sep 21;10(18):e022288. doi: 10.1161/JAHA.121.022288. Epub 2021 Sep 13. PMID 34514815

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The initial target was to randomize 3183 patients. This study was prematurely terminated (due to the neutral read-out of study RELAX-AHF-2) after 2666 patients were randomized. 16 patients had not qualified for randomization but were inadvertently randomized. These 16 patients did not enter the treatment phase and were not counted as started.
Period: Overall Study
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC)
Started (All Randomized Participants) | 1756 | 894
Full Analysis Set | 1756 | 894
Safety Set | 1729 (The Safety Set includes one patient not randomized but treated with serelaxin) | 894
Per Protocol Set | 1155 | 627
Completed | 1722 | 881
Not Completed | 34 | 13
Not completed — Lost to Follow-up | 14 | 8
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 14 | 3
Not completed — Technical Problems or Missing | 5 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC) | Total
Number analyzed (Participants) | 1756 | 894 | 2650
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.24 (10.349) | 75.95 (9.905) | 75.48 (10.205)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full Analysis Set
  Participants
    Female | 760 | 383 | 1143
    Male | 996 | 511 | 1507
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Full Analysis Set
  Participants
    Caucasian | 1706 | 869 | 2575
    Black | 4 | 4 | 8
    Asian | 5 | 2 | 7
    Unknown | 16 | 7 | 23
    Other | 25 | 12 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Worsening Heart Failure (WHF) / All Cause of Deaths Through Day 5
Description: In-hospital WHF through Day 5 post-randomization included worsening signs and/or symptoms of heart failure that required an intensification of intravenous therapy for heart failure or mechanical ventilation, renal or circulatory support. A central event adjudication committee was appointed to oversee the WHF primary endpoint adjudication.
Time Frame: 5 days
Population: Full Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 1756 | 894
Percentage of Participants | 4.95 | 6.94
Statistical Analysis 1: Comparison: Serelaxin + Standard of Care vs Standard of Care (SOC); Test type: Superiority; p = 0.0172, Gehan's generalized Wilcoxon test — One-sided p-value; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.51 to 0.98]

2. Secondary Outcome: Percentage of Participants With In-hospital Worsening Heart Failure/All-Cause Death/Readmission for Heart Failure Through Day 14
Description: WHF/death/readmission for heart failure through Day 14. WHF/deaths through Day 5 were adjudicated and confirmed by the Clinical Endpoint Committee, WHF/deaths after Day 5 through Day 14 and readmission through Day 14 were as reported by the investigators.
Time Frame: 14 days
Population: Full Analysis Set
Measure: Number; unit: Percentage of Patients
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 1756 | 894
Percentage of Patients | 8.49 | 10.63
Statistical Analysis 1: Comparison: Serelaxin + Standard of Care vs Standard of Care (SOC); Test type: Superiority; p = 0.0634, Gehan's generalized Wilcoxon test — Two-sided p-value; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.61 to 1.02]

3. Secondary Outcome: Percentage of Participants With Persistent Sign or Symptoms of Heart Failure / Non-Improvement at Any Post Baseline Visit Through Day 5
Description: Persistent or non-improvement in any signs or symptoms of HF at any post baseline visit up to Day 5.
Time Frame: 5 days
Population: Full Analysis Set (only evaluable patients with non-missing information included)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 1744 | 894
Percentage of Participants | 86 [84 to 87] | 91 [89 to 93]
Statistical Analysis 1: Comparison: Serelaxin + Standard of Care vs Standard of Care (SOC); Test type: Superiority; p < 0.0001, Chi-squared

4. Secondary Outcome: Percentage of Participants With Renal Deterioration at Any Post Baseline Visit Through Day 14
Description: Renal deterioration is defined as > or = 0.3 mg/dL increase from screening in serum creatinine.
Time Frame: 14 days
Population: Full Analysis Set (only evaluable patients with non-missing information included)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 1740 | 889
Percentage of Participants | 36 [34 to 38] | 44 [40 to 47]
Statistical Analysis 1: Comparison: Serelaxin + Standard of Care vs Standard of Care (SOC); Test type: Superiority; p = 0.0002, Chi-squared

5. Secondary Outcome: Length of Index Hospital Stay
Description: Length of stay (in hours) is defined as the index hospitalization discharge date and time minus the index hospitalization start date and time.
Time Frame: 30 Days
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 1756 | 894
hours | 251.28 (162.368) | 243.59 (160.270)
Statistical Analysis 1: Comparison: Serelaxin + Standard of Care vs Standard of Care (SOC); Test type: Superiority; p = 0.1392, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percentage of Participants With Adverse Events as Assessment of Safety and Tolerability of Serelaxin in AHF Patients
Time Frame: Adverse Events (AE): 5 Days / Serious Adverse Events (SAE): 14 days / All cause deaths 30 days
Population: Safety Set
Measure: Number; unit: Percentage of participants
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 1729 | 894
Percentage of participants
  Patients with any AE through Day 5 | 58.13 | 56.04
  Patients with any SAE through Day 14 | 12.38 | 11.97
  All cause deaths through Day 5 | 0.58 | 0.67
  All cause deaths through Day 14 | 1.91 | 2.01
  All cause deaths through Day 30 | 3.30 | 4.25

7. Secondary Outcome: Change From Baseline in Health-related Quality of Life Index Value, Assessed by EuroQoL EQ-5D-5L Questionnaire.
Description: EQ-5D-5L is a questionnaire designed to assess health status in adults consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The results were converted into a single index value using UK as the reference country for all countries. Range -0.3 (worst possible state) to 1 (best possible state).
Time Frame: Baseline, Day 5, Day 14
Population: Full Analysis Set (only evaluable patients with non-missing information included)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC)
Number analyzed (Participants) | 1545 | 793
units on a scale
  Day 5 | 0.28 (0.298) | 0.27 (0.292)
  Day 14: number analyzed (Participants) | 1486 | 756
  Day 14 | 0.32 (0.328) | 0.31 (0.317)
Statistical Analysis 1: Comparison: Serelaxin + Standard of Care vs Standard of Care (SOC); Day 5; Test type: Superiority; p = 0.3115, Mixed Models Analysis
Statistical Analysis 2: Comparison: Serelaxin + Standard of Care vs Standard of Care (SOC); Day 14; Test type: Superiority; p = 0.1236, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: All Cause Mortality: 30 days (additional deaths are included which occurred after the clinical trial reporting period of 30 days for up to 8 months post randomization); Serious Adverse Events: 14 days; Other non-serious Adverse Events (AEs): 5 days
Groups:
- Serelaxin + Standard of Care: Serelaxin (30 μg/kg/day) as continuous 48 hour intravenous infusion plus standard of care.
Arm/Group | Serelaxin + Standard of Care | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 63/1729 | 43/894
Serious Adverse Events (participants affected / at risk) | 214/1729 | 107/894
Other Adverse Events (participants affected / at risk) | 637/1729 | 324/894
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin + Standard of Care (N=1729) | Standard of Care (SOC) (N=894)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 6 | 4
Angina pectoris (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 4
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 3
Atrial fibrillation (Cardiac disorders) | 6 | 1
Atrioventricular block complete (Cardiac disorders) | 3 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 7 | 2
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 6 | 2
Cardiac failure (Cardiac disorders) | 38 | 26
Cardiac failure acute (Cardiac disorders) | 6 | 2
Cardiac failure chronic (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Cardiac hypertrophy (Cardiac disorders) | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 3 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 7 | 4
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 5 | 1
Myocardial infarction (Cardiac disorders) | 2 | 3
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 5 | 1
Ventricular tachycardia (Cardiac disorders) | 5 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 3 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Death (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 2
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Oropharyngitis fungal (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 11 | 6
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Skin bacterial infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 4
Urosepsis (Infections and infestations) | 2 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Heart rate decreased (Investigations) | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 0
Hypercapnic coma (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 4
Loss of consciousness (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Delirium (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 4
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 6 | 3
Renal impairment (Renal and urinary disorders) | 4 | 5
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Left atrial appendage occlusion (Surgical and medical procedures) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 7 | 2
Peripheral artery thrombosis (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serelaxin + Standard of Care (N=1729) | Standard of Care (SOC) (N=894)
Anaemia (Blood and lymphatic system disorders) | 49 | 9
Atrial fibrillation (Cardiac disorders) | 34 | 23
Cardiac failure (Cardiac disorders) | 81 | 56
Mitral valve incompetence (Cardiac disorders) | 28 | 12
Constipation (Gastrointestinal disorders) | 74 | 32
Diarrhoea (Gastrointestinal disorders) | 29 | 21
Nausea (Gastrointestinal disorders) | 40 | 17
Pyrexia (General disorders) | 24 | 21
Bronchitis (Infections and infestations) | 24 | 14
Urinary tract infection (Infections and infestations) | 56 | 26
Blood pressure systolic decreased (Investigations) | 49 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 47 | 35
Hypokalaemia (Metabolism and nutrition disorders) | 119 | 73
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 33 | 8
Headache (Nervous system disorders) | 45 | 18
Anxiety (Psychiatric disorders) | 27 | 16
Insomnia (Psychiatric disorders) | 58 | 21
Renal failure (Renal and urinary disorders) | 18 | 18
Renal impairment (Renal and urinary disorders) | 30 | 18
Hypotension (Vascular disorders) | 48 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT02064868/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT02064868/SAP_001.pdf